CLINICAL TRIAL: NCT03589105
Title: An Open-Label, Single-Arm Phase IV Study To Assess Ocrelizumab Efficacy, Safety, And Impact On Patient Reported Outcomes (PROS) In Patients With Active Relapsing Multiple Sclerosis
Brief Title: A Study to Provide Complementary Efficacy, Safety and Patient Reported Outcomes Data in Participants With Active Relapsing Forms of Multiple Sclerosis (MS) in a Pragmatic Setting
Acronym: PRO-MSACTIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML40359; 2018-000780-91 (EudraCT Number)
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ocrelizumab Treatment Cycles (Experimental): Each participant will receive an initial dose of two 300 mg infusions of Ocrelizumab each separated by 14 days followed by one single dose of 600 mg 24 weeks after the initial dose.
  Interventions: Drug: Ocrelizumab 300 mg; Drug: Ocrelizumab 600 mg

INTERVENTIONS:
Drug: Ocrelizumab 300 mg — Two doses of 300 mg infusion administered 14 days apart.
Drug: Ocrelizumab 600 mg — A single does of 600 mg infusion administered 24 weeks after the initial dose.

SUMMARY:
This national, open-label study is designed to give complementary efficacy, safety and patient reported outcomes (PROs) data in participants with active relapsing forms of MS. Participants will receive a maximum of 2 treatment cycles of ocrelizumab infusions: an initial dose of two 300 milligram (mg) infusions separated by 14 days followed by one single infusion of 600 mg ocrelizumab 24 weeks after the first infusion. Disease activity is determined by clinical relapses and/or Magnetic Resonance Imaging (MRI) activity.

ELIGIBILITY:
Inclusion Criteria:

* Age >/=18 years at screening
* Patients with relapsing forms of multiple sclerosis (RMS) with active disease defined by clinical or imaging features: (i) at least one clinical relapse over a 6-month period prior to screening; (ii) AND/OR at least one T1 gadolinium-enhancing lesion or new and/or enlarging T2 lesion as detected by brain Magnetic Resonance Imaging (MRI) performed over a 3 months period prior to screening with no change of Disease-Modifying Treatment(s) (DMT) compared to a previous MRI performed within 24 months before screening
* For women of childbearing potential: agreement to use an acceptable birth control method during the treatment period and for at least 12 months after the last dose of ocrelizumab
* Participants should be beneficiary of healthcare coverage under the social security system

Exclusion Criteria:

* Diagnosis of primary progressive MS
* Inability to complete an MRI (contraindications for MRI include but are not restricted to weight ≥140 kg, pacemaker, cochlear implants, presence of foreign substances in the eye, intracranial vascular clips, surgery within 6 weeks of entry into the study, coronary stent implanted within 8 weeks prior to the time of the intended MRI, etc…)
* Gadolinium intolerance
* History of ischemic cerebrovascular disorders (e.g., stroke, transient ischemic attack) or ischemia of the spinal cord
* History or known presence of central nervous system (CNS) or spinal cord tumor (e.g., meningioma, glioma)
* History or known presence of potential metabolic causes of myelopathy (e.g., untreated vitamin B12 deficiency)
* History or known presence of infectious causes of myelopathy (e.g., syphilis, Lyme disease, human T-lymphotropic virus 1 (HTLV-1), herpes zoster myelopathy)
* History of genetically inherited progressive CNS degenerative disorder (e.g., hereditary paraparesis; MELAS [mitochondrial myopathy, encephalopathy, lactic acidosis, stroke] syndrome)
* Neuromyelitis optica
* History or known presence of systemic autoimmune disorders potentially causing progressive neurologic disease (e.g., lupus, anti-phospholipid antibody syndrome, Sjogren's syndrome, Behçet's disease, sarcoidosis)
* History of severe, clinically significant brain or spinal cord trauma (e.g., cerebral contusion, spinal cord compression)
* Vulnerable patients (Patient referred to in Articles L. 1121-5 to L. 1121-8 and L. 1122-1-2 of the French Public Health Code)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Percentage of participants free of disease activity | From Enrollment to Week 48
  This outcome measure evaluates the impact of ocrelizumab on disease activity in participants with active Relapsing Multiple Sclerosis (RMS). Freedom of disease activity is defined as participant without any relapse from enrollment to Week 48 and without T1 Gadolinium-enhancing lesion detected by brain MRI at Week 48 and without any new and/or enlarging T2 lesion detected by brain MRI at Week 48.

SECONDARY OUTCOMES:
Annualized relapse rate | At Week 48
  Annualized relapse rate is defined as the total number of clinical relapses divided by the number of participant-years of study treatment exposure. This outcome measure describes the efficacy of ocrelizumab in active RMS participants.
Percentage of participants with stable, improved, or worsened expanded disability status scale (EDSS) | From Enrollment to Week 48
  This outcome measure describes the efficacy of ocrelizumab in active RMS participants.
Percentage of participants with confirmed disability progression at Week 24 (CDP24) | At Week 48
  This outcome measure describes the efficacy of ocrelizumab in active RMS participants.
Mean Change in EDSS | From Baseline to Week 48
  This outcome measure describes the efficacy of ocrelizumab in active RMS participants.
Percentage of relapse-free RMS participants | From Enrollment to Week 24 and Week 48
  This outcome measure describes the efficacy of ocrelizumab in active RMS participants.
Percentage of participants with no T1 gadolinium-enhancing lesion and no new and/or enlarging T2 lesion as detected by brain MRI | At Week 48
  This outcome measure describes the efficacy of ocrelizumab in active RMS participants.
Percentage of participants with no T1 gadolinium-enhancing lesion as detected by brain MRI | At Week 48
  This outcome measure describes the efficacy of ocrelizumab in active RMS participants.
Percentage of participants with no new and/or enlarging T2 lesion as detected by brain MRI | At Week 48
  This outcome measure evaluates the impact of ocrelizumab on disease activity in participants with active RMS.
Change in the score of MS symptom severity scale (SymptoMScreen) | At Week 24 and Week 48
  This outcome measure describes the impact of ocrelizumab on patient reported outcomes (MS symptom severity, fatigue, health-related quality of life with standard and disease specific scales, work productivity, and treatment satisfaction) in active RMS patients.
Change in the score of Modified Fatigue Impact Scale (MFIS) | At Week 24 and Week 48
  This outcome measure describes the impact of ocrelizumab on patient reported outcomes (MS symptom severity, fatigue, health-related quality of life with standard and disease specific scales, work productivity, and treatment satisfaction) in active RMS patients.
Change in the score of EuroQol 5-Dimension Questionnaire (EQ-5D-5L with Visual Analogue Scale (VAS)) for health-related quality of life | At Week 24 and Week 48
  This outcome measure describes the impact of ocrelizumab on patient reported outcomes (MS symptom severity, fatigue, health-related quality of life with standard and disease specific scales, work productivity, and treatment satisfaction) in active RMS patients.
Change in the score of Work Productivity and Activity Impairment scale (WPAI:SHP) | At Week 24 and Week 48
  This outcome measure describes the impact of ocrelizumab on patient reported outcomes (MS symptom severity, fatigue, health-related quality of life with standard and disease specific scales, work productivity, and treatment satisfaction) in active RMS patients.
Change in the score of Multiple Sclerosis International Quality Of Life Questionnaire (MusiQOL) | At Week 24 and Week 48
  This outcome measure describes the impact of ocrelizumab on patient reported outcomes (MS symptom severity, fatigue, health-related quality of life with standard and disease specific scales, work productivity, and treatment satisfaction) in active RMS patients.
Change in the score of Treatment Satisfaction Questionnaire for Medication (TSQM-14) | At Week 24 and Week 48
  This outcome measure describes the impact of ocrelizumab on patient reported outcomes (MS symptom severity, fatigue, health-related quality of life with standard and disease specific scales, work productivity, and treatment satisfaction) in active RMS patients.
Percentage of Participants with Adverse Events (AE) | From Baseline to Week 48
  This outcome measure describes ocrelizumab safety in active RMS patients. Severity of AEs is determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (46):
- France (46):
  - Centre hospitalier d'Agen; Neurologie, Agen
  - CHU Amiens Hopital Sud; Neurologie, Amiens Cedex1
  - CHU Angers, Batiement Larrey 2, Neurologie, Angers
  - CHU de Besancon Hopital Jean Minjoz; Service de Neurologie, Besançon
  - Groupe Hospitalier Pellegrin; Service de neurochirurgie B, Bordeaux
  - CHU Brest Hopital La Cavale Blanche; Neurologie, Brest
  - Hopital Pierre Wertheimer; Neurologie D, Bron
  - Hopital Cote De Nacre; Unite Neurologie Generale, Caen
  - CH Jean Rougier; Neurologie, Cahors
  - Ch De Calais; Hopital De Jour, Calais
  - CHMS Site Chambery; Neurologie, Chambéry
  - CHU Hopital Gabriel Montpied; Service de Neurologie, Clermont-Ferrand
  - Hôpital General - Service de neurologie; Service de neurologie, Dijon
  - CH de Gonesse; Neurologie, Gonesse
  - CHU de Grenoble; Neurologie, La Tronche
  - Centre hospitalier Andre Mignot; Neurologie, Le Chesnay
  - CH Le Mans; Neurologie, Le Mans
  - Centre hospitalier de Libourne Hopital Robert Boulin; Neurologie, Libourne
  - CH St Vincent de Paul, Lille
  - Hopital Roger Salengro; Service de Neurologie, Lille
  - CHU Dupruytren - Limoges; Neurologie, Limoges
  - Hopital européen de Marseille; Neurologie, Marseille
  - CHU de la Timone - Hopital d Adultes; Service de Neurologie, Marseille
  - Fondation Hopital Saint Joseph; Neurologie, Marseille
  - Gh De Meaux; Neurologie, Meaux
  - Centre hospitalier Annecy Genevois Site St Julien; Neurologie, Metz-Tessy
  - Centre hospitalier de Montlucon; Neurologie, Montluçon
  - Hopital Gui de Chauliac; Neurologie, Montpellier
  - Centre hospitalier de Mulhouse Hopital Emile Muller; Neurologie, Mulhouse
  - Hopital Central - CHU de Nancy; Service de Neurologie, Nancy
  - Hôpital Guillaume et René Laënnec; Service Neurologie, Nantes
  - Hôpital Pasteur; Service de Neurologie, Nice
  - CHU de Nîmes Hopital Caremeau; Service de Neurologie, Nîmes
  - Groupe Hospitalier Paris Saint Joseph; Service de Neurologie et Neurovasculaire, Paris
  - Fondation Rothschild; Service de Neurologie, Paris
  - Hopital Saint Antoine; Neurologie, Paris
  - CHU Poitiers - La Milétrie; Neurologie, Poitiers
  - Centre Hospitalier de Cornouaille; Neurologie, Quimper
  - Hopital Pontchaillou, Rennes
  - Hôpital Charles Nicolle; Service de Neurologie, Rouen
  - CHU Saint Etienne - Hôpital Nord; Neurologie, Saint-Priest-en-Jarez
  - Hopital Civil de Strasbourg; Service de Neurologie, Strasbourg
  - Hopital Foch; Neurologie, Suresnes
  - HIA de Toulon hôpital militaire; Neurologie, Toulon
  - Centre hospitalier Guy Chatiliez de Tourcoing; Neurologie, Tourcoing
  - Centre hospitalier de Valence; Neurologie, Valence

REFERENCES:
- [Derived] Pau D, Lotz M, Grandclaude G, Jegou R, Civet A. Interactive statistical monitoring to optimize review of potential clinical trial issues during study conduct. Contemp Clin Trials Commun. 2023 Mar 17;33:101101. doi: 10.1016/j.conctc.2023.101101. eCollection 2023 Jun. PMID 37008796
- [Derived] Manchon E, Laplaud D, Vukusic S, Labauge P, Moreau T, Kobelt G, Grouin JM, Lotz M, Pau D, Christine LF. Efficacy, safety and patient reported outcomes in patients with active relapsing multiple sclerosis treated with ocrelizumab: Final results from the PRO-MSACTIVE study. Mult Scler Relat Disord. 2022 Dec;68:104109. doi: 10.1016/j.msard.2022.104109. Epub 2022 Aug 13. PMID 36007299